CLINICAL TRIAL: NCT01923025
Title: A Single Centre, Open Label Study to Characterize the PK-PDE10A Enzyme Occupancy Relationship of RO5545965 After a Single Dose in Healthy Male Volunteers Using [11C]IMA107 Positron Emission Tomography
Brief Title: A PET Study With RO5545965 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BP28844; 2013-000538-36 (EudraCT Number)
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

ARMS (1):
- RO5545965 (Experimental)
  Interventions: Drug: RO5545965

INTERVENTIONS:
Drug: RO5545965 — Single dose

SUMMARY:
This single center, open-label study will evaluate the PK-PDE10A Enzyme Occupancy Relationship of RO5545965 after a single dose in healthy male volunteers by positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 25 to 50 years of age, inclusive; healthy status is defined by absence of evidence of any active or chronic disease
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Male subjects with female partners of child-bearing potential must use two methods of contraception, one of which must be a barrier method (i.e. condom), for the duration of the study and for 30 days after the last dose

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, haematological or allergic disease, metabolic disorder, cancer or cirrhosis
* History of clinically significant hypersensitivity or allergic drug reactions
* Any suspicion or history of alcohol abuse and/or consumption of other drugs of abuse
* Regular smoker (> 5 cigarettes, > 1 pipeful or > 1 cigar per day)
* Positive for hepatitis B, hepatitis C, or HIV infection
* Evidence of significant cardiovascular disease or disorder
* Participation in an investigational drug or device study within 3 months prior to first administration of the study drug or within 6 times the elimination half-life, whichever is longer
* Previous inclusion in a research and/or medical protocol or any clinical procedures involving nuclear medicine, PET, occupational exposure to ionizing radiation or radiological investigations with significant exposure to radiation, excluding dental X-ray and common X-rays of chest or extremities
* Subject has any condition that would prevent an MRI from accurately or safely being performed [eg, claustrophobia, cardiac pacemaker, metallic implants or clips]
* Subject unable to lie on his back in the PET or MRI scanner for a period of 90 minutes
* Contraindication for arterial cannulation
* Unsuitable veins for repeated venipuncture

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Brain PDE10 occupancy by RO5545965 | up to Day 2
PK/PD: Brain PDE10 inhibition in relationship to RO5545965 plasma concentrations | up to Day 2

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | up to 12 days
Pharmacokinetics: Plasma concentrations of RO5545965 | up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- London, United Kingdom